CLINICAL TRIAL: NCT04102735
Title: UNDER the Nose vs. Over the Nose Face Mask to Prevent Facial PRESSURE Ulcers During Face Mask-noninvasive Ventilation for Acute Hypercapnic Respiratory Failure
Brief Title: Under the Nose Face Mask to Prevent Facial Pressure Ulcers During NIV for Acute Hypercapnic Respiratory Failure (AHRF)
Acronym: UNDER PRESSURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Arras (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017-02
Record Dates: First submitted 2019-05-17; First posted 2019-09-25 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Acute Hypercapnic Respiratory Failure
Keywords: facial pressure ulcers; noninvasive ventilation; acute hypercapnic respiratory failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Over-the-nose facemask (Active Comparator): The AF541 oro-nasal mask is used with the over-the-nose mask cushion.
  Interventions: Device: Over-the-nose facemask
- Under-the-nose facemask (Experimental): The AF541 oro-nasal mask is used with the under-the-nose mask cushion.
  Interventions: Device: Under-the-nose facemask

INTERVENTIONS:
Device: Under-the-nose facemask — Patients with acute hypercapnic respiratory failure that need noninvasive ventilation and are randomized in the experimental group will receive the AF541 facemask used with the under-the-nose cushion.
  Arms: Under-the-nose facemask
Device: Over-the-nose facemask — Patients with acute hypercapnic respiratory failure that need non-invasive ventilation and are randomized in the comparator group will receive the AF541 facemask used with the over-the-nose cushion.
  Arms: Over-the-nose facemask

SUMMARY:
Noninvasive ventilation (NIV) is essential to treat acute hypercapnic respiratory failure. However, facial pressure ulcers appearing during facemask-delivered noninvasive ventilation are a source of NIV failure by interface intolerance.

A Philips facemask (model : AF541 SE Oro-Nasal mask) has the particularity to display two options for its positioning : a usually used "over-the-nose" positioning or an "under-the-nose" positioning that is supposed to reduce the incidence of facial pressure ulcers while keeping in the same time the qualities of a standard facemask.

The goal of this controlled randomized trial is to test the hypothesis that the "under-the-nose" positioning actually reduces the incidence of facial pressure ulcers, compared to the usually used "over-the-nose" positioning.

Results of this trial should lead to the proposition of a new interface strategy to prevent facial pressure ulcers and therefore to improve the tolerance of NIV via the use of facemasks displaying an "under-the-nose" positioning.

ELIGIBILITY:
Inclusion Criteria:

* Acute hypercapnic respiratory failure
* Initiation of NIV
* Estimated cumulative time of NIV upper than 12 hours for the first 48 hours of hospitalization

Exclusion Criteria:

* Contraindication for NIV (respiratory arrest, impossibility to fit the mask)
* Intubated patient
* Patient with a tracheostomy
* Post-extubation respiratory failure
* Patient exhibiting facial ulcers or skin lesions located at the insertion points of the mask before its hospitalization
* Person declining NIV
* Pregnancy
* Dying person

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2021-10-03 (Actual); Study Completion 2021-10-03 (Actual)

PRIMARY OUTCOMES:
Change of the incidence of facial pressure ulcers in the experimental arm compared to the control arm, within the first 3 days after NIV initiation. | 3 days after NIV initiation
  The primary endpoint is the development of a facial pressure ulcer within the first 3 days after NIV initiation

SECONDARY OUTCOMES:
Change of the delay for facial pressure ulcers to appear in the experimental arm, compared to the control arm | 7 days after NIV initiation
  This secondary endpoint is the delay (in hours) between NIV initiation and the development of a facial pressure ulcer.
Change of the severity of facial pressure ulcers in the experimental arm, compared to the control arm | 7 days after NIV initiation
  This secondary endpoint is the highest facial pressure ulcer severity score observed during patient hospitalization. This score is evaluated according to the National Pressure Ulcer Advisory Panel guidelines (Edsberg LE et al., 2016). Stage 1 pressure injury (the less severe score) corresponds to intact skin with a localized area of nonblanchable erythema. Stage 2 pressure injury corresponds to partial-thickness skin loss with exposed dermis. Stage 3 pressure injury corresponds to full-thickness skin loss. Stage 4 pressure injury (the most severe score) corresponds to full-thickness skin and tissue loss.
Change of the patient comfort in the experimental arm, compared to the control arm | 24 hours after NIV initiation
  This secondary endpoint is the comfort patient score at 24 hours after NIV initiation. This score is a numeric scale, validated for NIV (Lemyze M et al., 2013 ; Gregoretti C et al., 2002), going from 1 to 5 (1: very uncomfortable ; 2: uncomfortable ; 3: acceptable ; 4: quite comfortable ; 5: comfortable).
Change of the incidence of mask changes related to interface intolerance in the experimental arm, compared to the control arm | 7 days after NIV initiation
  This secondary endpoint is the incidence of mask changes related to interface intolerance during patient hospitalization.
Change of the incidence of NIV failure in the experimental arm, compared to the control arm | 7 days after NIV initiation
  This secondary endpoint is the incidence of NIV failure defined as the need to resort to intubation or palliative care (in the case of a do-not-intubate order) during patient hospitalization. NIV failures may be caused by refractory respiratory acidosis, refractory hypoxemia, pressure ulcers, interface intolerance, excessive unintentional air leaks or shock.

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm LEMYZE, MD, Principal Investigator — Centre Hospitalier Arras
Locations (2):
- France (2):
  - Centre Hospitalier Arras, Arras
  - Centre Hospitalier Lens, Lens

REFERENCES:
- [Background] Edsberg LE, Black JM, Goldberg M, McNichol L, Moore L, Sieggreen M. Revised National Pressure Ulcer Advisory Panel Pressure Injury Staging System: Revised Pressure Injury Staging System. J Wound Ostomy Continence Nurs. 2016 Nov/Dec;43(6):585-597. doi: 10.1097/WON.0000000000000281. PMID 27749790
- [Background] Lemyze M, Mallat J, Nigeon O, Barrailler S, Pepy F, Gasan G, Vangrunderbeeck N, Grosset P, Tronchon L, Thevenin D. Rescue therapy by switching to total face mask after failure of face mask-delivered noninvasive ventilation in do-not-intubate patients in acute respiratory failure. Crit Care Med. 2013 Feb;41(2):481-8. doi: 10.1097/CCM.0b013e31826ab4af. PMID 23263582
- [Background] Gregoretti C, Confalonieri M, Navalesi P, Squadrone V, Frigerio P, Beltrame F, Carbone G, Conti G, Gamna F, Nava S, Calderini E, Skrobik Y, Antonelli M. Evaluation of patient skin breakdown and comfort with a new face mask for non-invasive ventilation: a multi-center study. Intensive Care Med. 2002 Mar;28(3):278-84. doi: 10.1007/s00134-002-1208-7. Epub 2002 Feb 6. PMID 11904656
- [Derived] Lemyze M, Mallat J, Vangrunderbeek N, Granier M. Under-The-Nose Versus Over-The-Nose Face Mask to Prevent Facial Pressure Sores During Face Mask-Delivered Noninvasive Ventilation for Acute Hypercapnic Respiratory Failure: A Randomized Controlled Trial. Crit Care Med. 2023 Sep 1;51(9):1177-1184. doi: 10.1097/CCM.0000000000005902. Epub 2023 May 11. PMID 37166242